CLINICAL TRIAL: NCT05058209
Title: Effect of ZILRETTA Versus CELESTONE on Quality of Life, Pain, Neuromuscular Function, and Physical Performance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ROC Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1657878
Record Dates: First submitted 2021-09-07; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Triamcinolone; betamethasone sodium phosphate; Betamethasone

STUDY DESIGN:
Intervention Model Description: Randomized and Controlled Blinded Clinical Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Investigator and participant were blinded to study arm until the end of thier final visit/phone call. Medical assistant prepping injections and CCRC were not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Active Comparator): Triamcinolone acetonide extended-release injectable suspension. Single intra-articular extended-release injection of triamcinolone acetonide, to deliver 32 mg (5 mL). For intra-articular use only and should not be administered by the following routes: epidural, intrathecal, intravenous, intraocular, intramuscular, intradermal, subcutaneous.
  Interventions: Drug: Triamcinolone acetonide extended-release injectable suspension
- Arm 2 (Active Comparator): Betamethasone sodium phosphate and betamethasone acetate Injectable Suspension, USP 6 mg per mL, 3 mg per milliliter betamethasone, as betamethasone sodium phosphate, and 3 mg per milliliter betamethasone acetate. When oral therapy is not feasible, the Injectable Suspension is indicated for intramuscular use only.
  Interventions: Drug: Betamethasone sodium phosphate and betamethasone acetate Injectable Suspension

INTERVENTIONS:
Drug: Triamcinolone acetonide extended-release injectable suspension — Zilretta (Triamcinolone acetonide extended-release injectable suspension) is indicated as an intra-articular injection for the management of pain due to knee OA. The most commonly reported adverse reactions (incidence ≥1%) in clinical studies included sinusitis (2%), cough (2%), contusions (2%) and joint swelling (3%). For additional details, please see Package Insert (http://www.zilrettalabel.com/PI.pdf). The website for Zilretta additionally lists: joint pain, headache, back pain, sore throat and runny nose, and bruising as common side effects of receiving a Zilretta injection.
  Other Names: Zilretta
  Arms: Arm 1
Drug: Betamethasone sodium phosphate and betamethasone acetate Injectable Suspension — Celestone (betamethasone sodium phosphate and betamethasone acetate Injectable Suspension, USP 6 mg per mL) is indicated as an intra-articular injection for the management of chronic or long-term inflammation associated with multiple conditions including severe allergies, dermatological diseases, endocrine disorders, gastrointestinal diseases, hematologic disorders, neoplastic diseases, nervous system disorders, ophthalmologic diseases, renal diseases, respiratory diseases and rheumatic disorders, and others that may not be listed. Celestone Soluspan is available in generic form. The most commonly reported adverse reactions include acne, increased hunger, and weight gain.
  Other Names: Celestone
  Arms: Arm 2

SUMMARY:
The purpose of this study is to examine the pre, post, and follow up effects of a single ZILRETTA knee injection vs a single CELESTONE SOLUSPAN knee injection on physiological measure of self-reported quality of life, pain, physical function, and physical performance in individuals with osteoarthritis (OA) knee pain. The Primary Investigator (PI) will recruit 20 symptomatic knee OA patients for this study. Patients will be randomized into one of two treatment arms, Arm 1 (ZILRETTA injection) or Arm 2 (CELESTONE SOLUSPAN injection). Patients in Arm 1 will receive a single 5 mL IV injection of 32 mg ZILRETTA into the affected knee joint. Patients in Arm 2 will receive a 5ml IV injection of 6mg/ml CELESTONE SOLUSPAN into the affected knee joint. Each study arm will include 10 patients. All data will be collected prior to injection (baseline), as well as at 6-week (post 1) and 12-week follow-ups (post 2). Patients will blinded to treatment arm until after they complete their 12-week follow up.

DETAILED DESCRIPTION:
Individuals with knee osteoarthritis (OA) often experience pain and difficulty completing many everyday activities, such as walking or climbing stairs. It is a major cause of lost work time and a serious disability for many people. Although there is no cure for arthritis, there are many treatment options available to help manage pain and keep people active.

The ZILRETTA knee injection and CELESTONE knee injection are both FDA approved, extended-release corticosteroid, and are both common nonsurgical treatment options for patients with OA. Currently, there are no studies that have compared ZILRETTA and CELESTONE SOLUSPAN.

c. Aims Specific Aim 1: To determine the difference between intra-articular (IA) injection of Zilretta and intra-articular injection of Celestone in patients with knee OA improves physical performance (OARSI recommended physical performance measures).

Primary Hypothesis 1: Patients who receive knee IA injection of Zilretta or Celestone experience improved physical performance detectable at 6 weeks and 12 weeks.

Specific Aim 2: To determine the difference between IA injection of Zilretta and IA injection of Celestone in patients with knee OA improves physical function (KOOS-PF).

Hypothesis 2: Patients who receive knee IA injection of Zilretta or Celestone report improved patient-reported physical function (KOOS-PS) at 6 weeks and 12 weeks.

Specific Aim 3: To determine the difference between knee IA injection of Zilretta or Celestone in patients with knee OA improves quality of life (KOOS-QoL).

Hypothesis 3: Patients who receive knee IA injection of Zilretta or Celestone report improved quality of life (KOOS-QoL) detectable at 6 weeks and 12 weeks.

Specific Aim 4: To determine the difference between knee IA injection of Zilretta or Celestone in patients with knee OA improves pain based on numeric pain rating scale.

Hypothesis 3: Patients who receive knee IA injection of Zilretta or Celestone report improved pain level detectable at 6 weeks and 12 weeks.

II. Research Plan and Design

1. Study Objective The goal of this study is to evaluate the efficacy of Zilretta compared to Celestone for improving quality of life, pain, neuromuscular function, and physical performance.
2. Study Design The proposed study will compare Zilretta and Celestone effectiveness on patient-reported outcomes (quality of life, neuromuscular functioning, and pain) and physical performance (30-second chair standing test, 40m fast-paced walking test, stair ascent) related to knee arthritis. Patients will be chosen based on the level of arthritis of the knee and interest in non-surgical treatment options. After informed consent but before injection, Patients will be randomized into Zilretta or Celestone treatment arms. Patients will be consented and seen at baseline, in clinic at 6-weeks, and phone call follow-up at 12-weeks. Demographic information as well as any comorbidity or adverse events related to poor healing will be recorded.

Baseline

After completing informed consent but prior to injection, patients will complete:

* OARSI recommended physical performance tests (30-second chair standing test, 40m fast-paced walking test, stair ascent)
* KOOS-PS (Physical Function Shortform) - 7 questions
* KOOS-Quality of life subscale (QoL) - 4 questions
* Numerical Rating Scale (NRS) 6-week (Post 1)

During the 6-week follow up visit with the PI, patients will complete:

* OARSI recommended physical performance tests (30-second chair standing test, 40m fast-paced walking test, stair ascent) 12 weeks after treatment
* KOOS-PS (Physical Function Shortform) - 7 questions
* KOOS-Quality of life subscale (QoL) - 4 questions
* Numerical Rating Scale (NRS) 12-week (Post 2)

At 12-weeks post-injection, the Clinical Research Coordinator (CCRC) or Research Assistant (RA) will call each patient and patients will complete:

* KOOS-PS (Physical Function Shortform) - 7 questions
* KOOS-Quality of life subscale (QoL) - 4 questions
* Numerical Rating Scale (NRS)

If patients indicate any adverse events, high levels of pain, or have medical questions, the CCRC or RA will schedule the patient to be seen by the PI.

ELIGIBILITY:
Inclusion Criteria

* Men and women age 18 years or older with symptomatic bilateral knee OA
* Symptomatic knee OA will be defined as the presence of a definite osteophyte or joint space narrowing (KL Grade ≥2) on posteroanterior (PA) fixed flexion knee radiographs in subjects limited by bilateral pain rated on a Numerical Rating Scale as ≥ 4/10 on more than half of the days over the past month. Radiographic change must be visible at standard image size, irrespective of capability to detect more subtle changes through digital enhancement.
* Bilateral knee symptoms for ≥ 3 months prior to screening
* Has undergone at least one prior conservative osteoarthritis treatment (e.g. Physical therapy, analgesics)
* Ambulatory
* Willing and able to comply with the study procedures and visit schedules and ability to follow verbal and written instructions.

Exclusion Criteria

* Current consumption of more than 14 alcoholic drinks per week
* Clinical signs and symptoms of active knee infection or crystal disease of either knee within 1 month of screening
* Diagnosed with rheumatoid arthritis, Reiter's syndrome, psoriatic arthritis, gout, ankylosing spondylitis, or arthritis secondary to other inflammatory diseases; HIV, viral hepatitis; chondrocalcinosis, Paget's disease, or villonodular synovitis
* Diagnosed with leukemia, known presence of metastatic malignant cells, or ongoing or planned chemotherapeutic treatment.
* A gout attack in the past 2 years.
* Diseases of the spine, hip or other lower extremity joints judged by the investigator to be contributing to the pain in either knee (i.e. sciatica, nerve pain, hip OA). Note: Patients with hip replacement in either hip may be enrolled provided there is sufficient pain relief after hip replacement that analgesics are not required.
* Untreated symptomatic injury of either knee (e.g., acute traumatic injury, anterior cruciate ligament injury, clinically symptomatic meniscus injury characterized by a mechanical issue such as locking or catching).
* Uncontrolled diabetes (HbA1c >7.2)
* Women who report pregnancy or childbearing potential and not using acceptable contraceptive measures (oral contraceptive, long acting reversible contraceptive therapy) (due to the potential for change in body mass and distribution to alter knee symptoms over the period of follow-up).
* Presence of surgical hardware or other foreign body intended to treat arthritis or cartilage-related pathology in either knee.
* Arthroscopy or open surgery of either knee within 6 months of screening.
* Planned/anticipated surgery of either knee during the study period.
* Use of systemic immunosuppressant within 6 weeks of screening.
* Oral corticosteroids (investigational or marketed) within 2 weeks of screening (unless on chronic stable dose for >3 months).
* IA corticosteroid (investigational or marketed) in either knee within 3 months of screening.
* IV or IM (Intramuscular) Corticosteroid injection (investigational or marketed) within 3 months of screening.
* Any other IA drug/biologic use within 6 months of screening or 5 half-lives (whichever is longer) (e.g., hyaluronic acid, platelet-rich plasma (PRP) injection, stem cells, prolotherapy and amniotic fluid injection).
* Any documented clinically significant degree of cognitive impairment or other condition, finding, or psychiatric illness at screening which, in the opinion of the investigator, could compromise subject safety.
* Any condition other than OA of the knee which, in the opinion of the investigator, affects the ability to ambulate to a sufficient degree to interfere with the assessment of the safety and treatment effects of the study injection.
* Participated in any interventional drug or device trial within 30 days prior to screening or concurrent participation in another research study that could complicate interpretation of the study findings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
OARSI - 30-second Chair Stand | Baseline (removed due to COVID)
  The maximum number of chair stand repetitions possible in a 30 second period (2-4).
OARSI - 30-second Chair Stand | 6 week (removed due to COVID)
  The maximum number of chair stand repetitions possible in a 30 second period (2-4).
OARSI - 30-second chair standing test | 12 week (removed due to COVID)
  The maximum number of chair stand repetitions possible in a 30 second period (2-4).
OARSI - 40m Fast Paced Walk | Baseline (removed due to COVID)
  A fast-paced walking test that is timed over 4 x 10m (33 ft) for a total 40 m (132 ft) (2).
OARSI - 40m Fast Paced Walk | 6 week (removed due to COVID)
  A fast-paced walking test that is timed over 4 x 10m (33 ft) for a total 40 m (132 ft) (2).
OARSI - 40m Fast Paced Walk | 12 week (removed due to COVID)
  A fast-paced walking test that is timed over 4 x 10m (33 ft) for a total 40 m (132 ft) (2).
OARSI - stair ascent | Baseline (removed due to COVID)
  The time (in seconds) it takes to ascend and descend a flight of stairs (2-6). The number of stairs will depend on individual environmental situations. Where possible, the 9-step stair test with 20cm (8 inch) step height and handrail is recommended.
OARSI - stair ascent | 6 week (removed due to COVID)
  The time (in seconds) it takes to ascend and descend a flight of stairs (2-6). The number of stairs will depend on individual environmental situations. Where possible, the 9-step stair test with 20cm (8 inch) step height and handrail is recommended.
OARSI - stair ascent | 12 week (removed due to COVID)
  The time (in seconds) it takes to ascend and descend a flight of stairs (2-6). The number of stairs will depend on individual environmental situations. Where possible, the 9-step stair test with 20cm (8 inch) step height and handrail is recommended.
KOOS-PS (Physical Function Shortform) | 6 week
  Scoring: Never/none=0, Monthly/mild=1, Weekly/moderate=2, Daily/severe=3, Always/extreme=4. Calculate the mean score for the 11 items, and divide by the maximum possible score for each item (i.e. 4). Traditionally in orthopedics, 100 indicates no problems and 0 indicates extreme problems.
  The normalized score is transformed to meet this standard. Please use the formula provided below. 100 - [(mean score PF1-PF11)/4 *100]
KOOS-PS (Physical Function Shortform) | Baseline
  Scoring: Never/none=0, Monthly/mild=1, Weekly/moderate=2, Daily/severe=3, Always/extreme=4. Calculate the mean score for the 11 items, and divide by the maximum possible score for each item (i.e. 4). Traditionally in orthopedics, 100 indicates no problems and 0 indicates extreme problems.
  The normalized score is transformed to meet this standard. Please use the formula provided below. 100 - [(mean score PF1-PF11)/4 *100]
KOOS-PS (Physical Function Shortform) | 12 week
  Scoring: Never/none=0, Monthly/mild=1, Weekly/moderate=2, Daily/severe=3, Always/extreme=4. Calculate the mean score for the 11 items, and divide by the maximum possible score for each item (i.e. 4). Traditionally in orthopedics, 100 indicates no problems and 0 indicates extreme problems.
  The normalized score is transformed to meet this standard. Please use the formula provided below. 100 - [(mean score PF1-PF11)/4 *100]
KOOS-Quality of life subscale (QoL) | Baseline
  The KOOS's five patient-relevant dimensions are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
KOOS-Quality of life subscale (QoL) | 6 week
  The KOOS's five patient-relevant dimensions are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
KOOS-Quality of life subscale (QoL) | 12 week
  The KOOS's five patient-relevant dimensions are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Numerical Rating Scale (NRS) | Baseline
  patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable
Numerical Rating Scale (NRS) | 6 week
  patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable
Numerical Rating Scale (NRS) | 12 week
  patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Sara C DePaoli, Study Director — ROC Foundation; Timothy J Bray, MD, Principal Investigator — ROC Foundation
Locations (1):
- Reno Orthopedic Center, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No